CLINICAL TRIAL: NCT00341692
Title: Pilot Study to Collect Normal Breast Tissue From Organ and Tissue Donors
Brief Title: Studying Normal Breast Tissue and Cancer Risk
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903158; 03-C-N158
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases
Keywords: Mammary; Development; Cancer; Risk; Genes
MeSH Terms: conditions — Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Samples of normal breast tissue: Samples of normal breast tissue from organ donors for assessment of histology.

SUMMARY:
Breast cancer is the most common cancer among women in the United States. Breast cancer research has been hampered by the difficulty in collecting normal breast tissue. In this study, researchers will obtain samples of normal breast tissue from organ donors and will collect risk-factor data from next-of-kin.

The purpose of this study is to learn how normal breast develops and responds to stresses that are known to increase a woman s chance of developing breast cancer.

Following the breast-tissue donation from 20 volunteers, surgical technicians will make small incisions in the skin and tissue of the breast and remove several samples measuring about one-inch. Technicians also will take samples of the uterine lining to estimate the date of the last menstrual period. The tissue will then be sent to the National Cancer Institute for laboratory research studies. Steps will be taken to ensure that the identity of the participants remains confidential.

DETAILED DESCRIPTION:
This pilot project, funded by a Breast Cancer Faculty Infrastructure Award, would determine the feasibility of obtaining samples of normal breast tissue from organ donors and collecting risk factor data from next-of-kin. The underlying goal of this initiative is to determine the associations between stages of breast development, risk factors for breast cancer, and gene expression. The study investigators are members of DCEG, CCR and the Transplant Resource Center of Maryland (TRC), a non-profit organization certified by HCFA and the state that processes most organ and tissue donations in Maryland. Trained staff or social workers employed by TRC who routinely obtain consent for donation from next-of-kin will also obtain consent for this study. The existing consent form for organ or tissue donation also includes informed consent for donation of tissue for research. Following organ procurement from 20 volunteers, trained surgical technicians employed by TRC who routinely assist intra-operatively, will sterilely remove tissue from each breast quadrant and split the samples; one portion will be embedded in OCT and snap frozen in liquid nitrogen and the other fixed in 10% buffered formalin. Samples of adipose tissue, blood, urine and endometrium (for menstrual dating) will also be obtained. MES in conjunction with SMH and BKV will assess the samples histopathologically and determine the quantity and quality of macromolecules (RNA, DNA, protein) contained within the tissues. Pending demonstration of the feasibility of this general approach, we will pursue additional funding for a larger study with optimized procedures. We have stopped recruiting patients.

ELIGIBILITY:
* INCLUSION CRITERIA

The study will enroll girls or women aged 11 years or older.

EXCLUSION CRITERIA

Men are excluded.

Ages: 11 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples of normal breast tissue from organ donors for assessment of histology.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2003-04-07 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Histological features | cross-sectional
  descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Benson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chuaqui RF, Bonner RF, Best CJ, Gillespie JW, Flaig MJ, Hewitt SM, Phillips JL, Krizman DB, Tangrea MA, Ahram M, Linehan WM, Knezevic V, Emmert-Buck MR. Post-analysis follow-up and validation of microarray experiments. Nat Genet. 2002 Dec;32 Suppl:509-14. doi: 10.1038/ng1034. PMID 12454646
- [Background] Kononen J, Bubendorf L, Kallioniemi A, Barlund M, Schraml P, Leighton S, Torhorst J, Mihatsch MJ, Sauter G, Kallioniemi OP. Tissue microarrays for high-throughput molecular profiling of tumor specimens. Nat Med. 1998 Jul;4(7):844-7. doi: 10.1038/nm0798-844. PMID 9662379
- [Background] Gruvberger S, Ringner M, Chen Y, Panavally S, Saal LH, Borg A, Ferno M, Peterson C, Meltzer PS. Estrogen receptor status in breast cancer is associated with remarkably distinct gene expression patterns. Cancer Res. 2001 Aug 15;61(16):5979-84. PMID 11507038